CLINICAL TRIAL: NCT03228199
Title: PROductivity Study of Presbyopia Elimination in Rural-dwellers (PROSPER)
Acronym: PROSPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Congdon Nathan (Other)
Collaborators: Queen's University, Belfast (Other); Clearly (Other); COMMUNITY EYE CARE FOUNDATION (CECF) (Unknown); Aravind Eye Care System (Other); University of British Columbia (Other); Amalgamated Plantations Private Limited (Unknown); VisionSpring (Other)
Responsible Party: Sponsor-Investigator, Congdon Nathan, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PROSPER (IRB - LNEH/88/2017)
Record Dates: First submitted 2017-06-03; First posted 2017-07-24 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Presbyopia
Keywords: Randomised Control Trial; Productivity; Agricultural workers; India; Vision correction
MeSH Terms: conditions — Presbyopia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomization, Balancing, and Intervention: Eligible workers completing baseline productivity assessment will be enrolled into the study, and assigned at random to one of the below groups:
  Intervention Group: Will immediately receive a free pair of presbyopic glasses through the Clear Vision Workplace program. These glasses will correct the worker's vision at their usual working distance by placing the vision chart on the top of a tea bush and directing the participant to stand as usual in picking tea. The gasses will not correct astigmatism. Distance refractive errors will be corrected for those with uncorrected VA < 6/12 in the better-seeing eye.
  Control Group: Will be deferred to receive free presbyopic spectacles after the 12 weeks evaluation period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Main outcome and masking: The daily mean weight of tea picked will be calculated for each worker for the 4 weeks baseline and for the 12 weeks evaluation period. The difference between these two means will be calculated for each worker, and the mean of this value will be calculated for each randomised group, with the main study outcome being the difference between these values for each group. It will not be practical to mask participants as to their study group assignment (the investigators do not feel that providing sham near correction of Plano power is ethical). However, the APPL staff measuring the weight and quality outcomes will be masked to a worker's group assignment by having an intermediate person receive the tea from the worker and carry it to the weighing station each day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presbyopic Glasses/ Intervention Group (Other): Immediate provision of a free pair of spherical presbyopic glasses to correct the worker's vision for optimal picking distance as measured using a chart placed at the top of a typical tea bush.
  Interventions: Other: Intervention group
- Control Group (Other): Will be deferred to receive spectacles as above, after the 12 weeks evaluation period.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention group — Will immediately receive a free pair of presbyopic glasses through the Clear Vision Workplace program. These glasses will correct the worker's vision at their usual working distance, and will not correct astigmatism.
  Arms: Presbyopic Glasses/ Intervention Group
Other: Control Group — Will be deferred to receive spectacles as above, after the 12 week evaluation period.
  Arms: Control Group

SUMMARY:
This trial seeks to establish, using a randomized, controlled design, the impact of near eyesight correction on the productivity of presbyopic agricultural workers in India, as measured by weight of tea picked.

DETAILED DESCRIPTION:
Main research question being addressed: To establish, using a randomized, controlled design, the impact of near eyesight correction on the productivity of presbyopic agricultural workers in India, as measured by weight of tea picked.

Primary outcomes to be measured: Change in mean daily weight of tea picked per worker during a 12 weeks period after randomisation compared to a 4 weeks baseline period prior to randomisation. (See details below under Main Outcome.)

I. Background: Importance of research topic, Particular Features of setting Uncorrected presbyopia is an expensive problem for the world. Lost productivity among adults who need eyeglasses has been estimated to cost the global economy $227 billion every year, [1,2] and illiteracy may lead to a further $3 trillion in annual global economic losses. It has been shown that 74% of illiterate adults failed one or more parts of a vision screening. [3] However, in order to motivate governments, industry and other key stakeholders to invest in solving the problem of uncorrected near vision in adults, higher-quality data on the productivity impact of correction are needed. Current studies are suggestive, but carefully-performed randomized trials are still lacking in the published literature.

An unpublished University of Michigan (USA) working paper found that correcting near-vision loss with glasses yields an increase in productivity of up to 34%, though no control group was included, and the outcome assessed was not precisely defined. An unpublished impact assessment conducted by Building Resources Across Communities (BRAC), the world's largest NGO in the number of staff, concluded that 90% of individuals experiencing near-vision loss in Bangladesh encountered problems with their daily work; and, on average, 23% reported that their income was compromised.[4] In Rwanda, Lifetime Consulting & Partners found that workers with poor vision who did not wear glasses were three times more likely to be asked by supervisors to repeat their work of sorting coffee beans than after receiving and wearing glasses.[4] Again, no control group was included, and this work has not been published. Furthermore, a Dalberg Global Development Advisors study of adults in India who had their vision corrected with glasses found that 65% reported an increase in independence in movement and travel, and 59% reported improved work productivity, [5] but these outcomes were not confirmed quantitatively or objectively. Finally, a population study of 1008 older adults in Shenyang, northern China, found that those with uncorrected presbyopia (69%) were more likely to report diminished accomplishment due to vision (P = 0.01, adjusted for age, sex, education, and distance vision) than were those without presbyopia. [6] The impact of correcting presbyopia was not studied in a prospective fashion.

In summary, available data are consistent with the idea that correcting presbyopia can lead to significant improvements in productivity among adult workers. However, in the absence of high-quality randomized trials, it is very difficult to be certain about cause and effect: it is equally plausible that the economic burden of poverty could result in failure to purchase glasses, rather than the reverse. Lack of control groups and carefully-defined productivity outcomes in many studies further hinder interpretation. Policy makers and industry partners require more convincing data in order to commit to the support of programs of vision correction.

Features of this setting:

A high proportion (> 50%) of workers have presbyopia in this large workforce, and previous projects by Vision Spring have shown that the large majority of these workers have no presbyopic correction.

The primary outcome (daily weight of tea picked) is measured and recorded by Amalgamated Tea as part of routine practice.

The work population is very stable, and data from previous years have been used for sample size calculations.

The project will be carried out during the high season (July through October) when the amount of tea picked is limited by the labourer and not by the growth of the plants. Further, these agricultural workers are strongly incentivized to pick more tea, because they are paid by weight, and thus gain in income when their personal productivity increases.

II. Experimental plan

Study design: Randomized, investigator-masked controlled trial

Methods to be used:

Population: Presbyopic (generally age >= 40 years) tea workers at the Amalgamated Plantations Pvt Ltd (APPL) in Assam, India.

Baseline data acquisition: Demographic and clinical: Age, sex, contact information, habitual and best-corrected visual acuity at near and distance; power of distance and near refractive error in each eye; workers with acuity not improving to 6/7.5 in either eye at distance will undergo dilated fundus examination and will be referred to a local collaborating facility for care if needed. Work productivity: Daily mean weight of tea picked during a 4 weeks baseline period prior to randomisation.

Recruitment and consent: Approximately 1500 APPL workers aged 40 years or more will undergo assessment of above clinical criteria ("Baseline data acquisition") by VisionSpring local staff, assisted by APPL as part of the on-going Clear Vision Workplace program. Those meeting inclusion criteria (see below) will be invited to join to the study and complete informed consent forms. Recruitment will continue until approximately 700 persons have joined the study (see sample size calculations below). Baseline work productivity will be measured as outlined above for a 4-week period).

Randomization, Balancing, and Intervention: Eligible workers completing baseline productivity assessment will be enrolled into the study, and assigned at random to one of the below groups:

Intervention Group: Will immediately receive a free pair of presbyopic glasses through the Clear Vision Workplace program. These glasses will correct the worker's vision at their own usual working distance (methodology described in the full protocol), and will not correct astigmatism. Distance refractive errors will be corrected for those with uncorrected VA < 6/12 in the better-seeing eye, but such persons will be excluded from the trial.

Control Group: Will be deferred to receive free presbyopic spectacles after the 12 weeks evaluation period.

Balance of the groups on age and baseline work productivity, will be assessed and maintained insofar as possible, and allocation concealment prior to randomisation will be ensured through the use of a secure process so that neither the participant nor the person recruiting them to the study will know in advance whether or not they will receive spectacles immediately or after 12 weeks.

Randomization methodology: Eligible workers completing baseline data collection will be enrolled into the study, and stratified into eight groups according to age (<50, >=50), sex and baseline work productivity (<median, >=median), then participants among each of the eight groups will be assigned at random to one of the study arms.

An independent statistician having no contact with participants will generate the randomization sequence using a computer system that is inaccessible until after recruitment. The participants in each stratified group will be assigned to either the intervention or control group in a 1:1 ratio with the block size of six. The participants will know their group assignment. However, the APPL staff measuring the weight and quality outcomes will be masked to a worker's group assignment by having an intermediate person receive the tea from the worker at the weighing station each day.

Main outcome and masking: The daily mean weight of tea picked will be calculated for each worker for the 4 weeks baseline and for the 12 weeks evaluation period. The difference between these two means will be calculated for each worker, and the mean of this value will be calculated for each randomised group, with the main study outcome being the difference between these values for each group. It will not be practical to mask participants to their study group assignment (the investigators do not feel that providing sham near correction of Plano power is ethical). However, the APPL staff measuring the weight outcomes will be masked to a worker's group assignment by having an intermediate person receive the tea from the worker and carry it to the weighing station each day. Secondary outcomes will include visual quality of life in both groups, self-reported wear of the study spectacles in the intervention group, self-reported purchase and use of glasses in the control group, independent compliance observations, quality of tea picked (if possible to assess) and the proportion of workers who work than less than 10 days in a month during the 12 weeks evaluation period.

Study hypothesis: Productivity gains in the Intervention Group will be significantly greater than those in the Control Group when the 12 weeks evaluation period is compared to the 4 weeks baseline period.

Sample size calculations: With two-sided significance level of P=0.05, power of 80%, a daily mean of 25.0 (SD: 5.0) kg of tea picked at baseline (among persons working >= 10 days in a month), and allowing for 20% loss to follow-up, a sample size of 160 persons (80 per group) will be sufficient to detect a 10% greater increase in daily mean weight of tea picked in the intervention group compared to the control group (primary outcome). However, in order to have sufficient data to conduct adequately powered analyses to compare the results for persons aged 40 years and above, with those for persons aged at least 45 years and at least 50 years, we will aim to recruit a total of 700 participants. These subgroup analyses will be important for informing future policy, for example, if choices need to be made about which, if any, age groups should be targeted for eyeglasses.

Statistical methods: The analysis of the primary outcome (as defined above) between randomised groups will be done with and without adjustment for potential determinants of productivity at baseline (including age and sex) and during the evaluation period (including self-reported use of glasses in the intervention group and self-reported purchase and use of glasses among the control group). The mean daily data for participants working <10 days in a month during the evaluation period will be excluded from the main analyses in sensitivity analyses to assess the impact of these workers on the overall results (both in relation to the effect estimate and its confidence interval). Main analysis will also include age-stratified analysis of participants (for example, 40-44, 45-49, 50-59, and 60 and above).

Study Roles and Monitoring: The principal investigator will be responsible for final approval of the study protocol, overall study coordination and completing the UK ethical review. The principal investigator has a long-standing working relationship with VisionSpring (VS) and extensive experience in design and execution of randomised trials on a refractive error in settings of limited resources. The principal investigator will visit India on two occasions: During the Study Preparation period and at the time of the Baseline examination. The VS India team will be responsible for coordinating fieldwork. VS has worked in India for 10 years, and with APPL since 2014, and has extensive experience in carrying out presbyopic screening and provision of near spectacles in India and a wide variety of LMIC settings. APPL will provide support for the baseline examination, administration of the intervention and the end line distribution of glasses to the Control Group. APPL will also be primarily responsible for the collection of the primary study outcome (mean daily weight of picked tea) and the secondary outcome of the quality of picked tea in both groups.

Dissemination strategy: The project management team will prepare a dissemination strategy which balances the requirements of academic audiences (peer-reviewed journal publications and conference presentations) with those of policy-makers and local patients and practitioners in both the UK and India and our NGO partners. In submitting findings to a range of academic journals, the investigators will focus on internationally-recognized journals with high impact, particularly those such as BMJ and Lancet Global Health with open access policies, making the papers more available to researchers and policy-makers in LMICs. The investigators will collaborate with the Cochrane Eyes and Vision group to help them update reviews on the economic impact of the correction of refractive error. At the conclusion of the main trial, principal results will be available in English and several Indian languages and in graphic format on a mobile-friendly project website. Results will also be shared through organizations such as our Indian research partners and various locally-active eye health NGOs.

Funding: Primary funding provided by Clearly (Clearly.World), free glasses provided by VisionSpring (VisionSpring.org).

ELIGIBILITY:
Inclusion Criteria:

* Employee of APPL for 1 year
* Aged >= 40 years
* Habitual near visual acuity of >= 0.8M (<=6/12) at 40cm in both eyes, correctable to <=0.5M (>=6/7.5) in both eyes with near glasses
* Uncorrected distance vision >= 6/7.5 in the better-seeing eye
* The participant worked and has data available on weight of tea picked for >=10 days in the previous 4 weeks (This will largely exclude men in this setting).
* Ability to give informed consent

Exclusion Criteria:

* Eye disease detected on baseline eye exam
* Current ownership of near correction capable of improving near visual acuity to <= 0.8M (>= 6/12) in either eye
* Unlikely to complete follow-up due to unsatisfactory work performance, plans to move out of the area, etc.
* Need for distance correction to achieve distance vision of >= 6/7.5 in the better-seeing eye.
* Inability to achieve best-corrected visual acuity with spherical power glasses only (that is: need for astigmatic correction to achieve best-corrected near visual acuity)

Persons with eye problems detected on the examination will be referred for definitive care at local facilities, and distance refractive errors will be corrected with free bifocals for those with uncorrected VA < 6/12 in the better-seeing eye.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
The impact of near correction of the vision on productivity of agricultural workers in India will be measured. | 4 to 5 months
  The main outcome will be change in mean daily weight of tea picked per worker during a 12 weeks period after randomisation to intervention or control, compared to a 4 weeks period prior to the randomisation.

SECONDARY OUTCOMES:
The impact of near correction of the vision on productivity of agricultural workers in India | 4 to 5 months
  Secondary outcomes will include visual quality of life in both groups, self-reported wear of the study spectacles in the intervention group, self-reported purchase and use of glasses in the control group, independent compliance observations and the proportion of workers who work less than 10 days in a month during the 12 weeks evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, Principal Investigator — Queen's University, Belfast
Locations (1):
- Amalgamated Plantations Private Limited (APPL), Tezpur, Assam, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fricke TR, Holden BA, Wilson DA, Schlenther G, Naidoo KS, Resnikoff S, Frick KD. Global cost of correcting vision impairment from uncorrected refractive error. Bull World Health Organ. 2012 Oct 1;90(10):728-38. doi: 10.2471/BLT.12.104034. Epub 2012 Jul 12. PMID 23109740
- [Result] Frick KD, Joy SM, Wilson DA, Naidoo KS, Holden BA. The Global Burden of Potential Productivity Loss from Uncorrected Presbyopia. Ophthalmology. 2015 Aug;122(8):1706-10. doi: 10.1016/j.ophtha.2015.04.014. PMID 26190438
- [Result] Johnson R, Zaba J. The link: Vision and illiteracy. J of Behav Optometry 1994;5:41-3
- [Result] EYEIliance, Eyeglasses for global development: Bridging the visual divide. June 2016 report
- [Result] Dalberg Global Development Advisors 2015. Impact study of Essilor's Eye Mitra optician programme in India (a programme of the Essilor Group's 2.5 New Vision Generation division)
- [Result] Lu Q, Congdon N, He X, Murthy GV, Yang A, He W. Quality of life and near vision impairment due to functional presbyopia among rural Chinese adults. Invest Ophthalmol Vis Sci. 2011 Jun 13;52(7):4118-23. doi: 10.1167/iovs.10-6353. PMID 21508106
- [Derived] Reddy PA, Congdon N, MacKenzie G, Gogate P, Wen Q, Jan C, Clarke M, Kassalow J, Gudwin E, O'Neill C, Jin L, Tang J, Bassett K, Cherwek DH, Ali R. Effect of providing near glasses on productivity among rural Indian tea workers with presbyopia (PROSPER): a randomised trial. Lancet Glob Health. 2018 Sep;6(9):e1019-e1027. doi: 10.1016/S2214-109X(18)30329-2. Epub 2018 Jul 23. PMID 30049615

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03228199/Prot_SAP_008.pdf